CLINICAL TRIAL: NCT06402981
Title: A Clinical Study on the Analysis of Risk Factors for the Occurrence of PD-1/PD-L1 Inhibitor-associated Liver Injury in Lung Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jiajia Chen, Chief Physician of the First Affiliated Hospital,Zhejiang University School of Medicine, Zhejiang University
Other Study IDs: IIT20240464A
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Immune Checkpoint Inhibitors; Liver Injury
Keywords: PD-1/PD-L1 inhibitor; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- liver damage group: Lung cancer patients using PD-1/PD-L1 inhibitors with hepatic injury as determined by the hepatic index criteria set by the Common Terminology Criteria for Adverse Events (CTCAE 5.0)
  Interventions: Other: High risk prediction model for liver injury
- No liver damage group: Lung cancer patients with PD-1/PD-L1 inhibitors who are judged not to have liver injury according to the liver index criteria set by the Common Terminology Criteria for Adverse Events (CTCAE 5.0)
  Interventions: Other: High risk prediction model for liver injury

INTERVENTIONS:
Other: High risk prediction model for liver injury — Risk Prediction Model for Liver Injury After Use of PD-1/PD-L1 Inhibitors

SUMMARY:
The goal of this observational study is to investigate the risk factors of PD-1/PD-L1 inhibitor-associated liver injury, to construct a prediction model for the occurrence of liver injury. The main questions it aims to answer are:

* Exploring risk factors for liver injury.
* Constructing a Predictive Model for the Occurrence of Liver Injury in PD-1/PD-L1 Inhibitor-Related Liver Injury.
* Improving immunotherapy protocols for lung cancer patients.

DETAILED DESCRIPTION:
PD-1/PD-L1 inhibitors have achieved surprising results in lung cancer treatment and have been approved by the FDA for the treatment of different types of lung cancer. Their overall toxicity is lower than that of standard chemotherapy, but a number of immune-related adverse events have been reported clinically. Liver injury is one of the leading causes of death from adverse events due to PD-1/PD-L1 inhibitors. The occurrence of immune-related liver damage has an important impact on the tumor treatment and prognosis of patients. Most of the current domestic and international studies focus on the overall description and study of PD-1/PD-L1 antibody-related adverse events, and there is no definitive description of the risk factors for the development of immune-related liver injury in lung cancer patients. The aim of this project is to review the clinical data of lung cancer patients treated with PD-1/PD-L1 inhibitors from 2020.01 to 2024.06, to investigate the risk factors of PD-1/PD-L1 inhibitor-associated liver injury, to construct a prediction model for the occurrence of liver injury, and to take measures to prevent the occurrence of fatal immune liver injury, which is of great significance to the immunotherapy of clinical tumor patients. It is of great significance to the immunotherapy of clinical tumor patients.

ELIGIBILITY:
Inclusion Criteria:

1. Lung cancer patients who have received at least one and more PD-1/PD-L1 inhibitor treatments;
2. Gender is not limited, age 18-80 years old

Exclusion Criteria:

1. Severe liver injury prior to immunotherapy (elevation of transaminases, alkaline phosphatase, and glutamyl aminotransferase more than 5 times the upper limit of normal).
2. Patients who, in the opinion of the investigator, are not suitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients treated with PD-1/PD-L1 inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
liver injury | 8 weeks
  The occurrence of immunosuppressant-associated liver damage was determined according to criteria set by the Common Terminology Criteria for Adverse Events (CTCAE 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Jiajia Chen, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No